CLINICAL TRIAL: NCT04094025
Title: A Randomized, Evaluator-blinded Study to Evaluate Skin Irritation and Sensitization of d-Amphetamine Transdermal System in Healthy Adults
Brief Title: Irritation and Sensitization Study of d-Amphetamine Transdermal System
Acronym: dATS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Noven Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: N25-018
Record Dates: First submitted 2019-09-11; First posted 2019-09-18 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2019-12

CONDITIONS: Cumulative Irritation and Sensitization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- dATS patch (Experimental): dATS, placebo and saline will be administered simultaneously
  Interventions: Drug: dATS

INTERVENTIONS:
Drug: dATS — d-Amphetamine Transdermal System

SUMMARY:
The study will assess skin irritation as well as sensitization for d-ATS patch in healthy subjects.

DETAILED DESCRIPTION:
This is a randomized, evaluator-blinded study consisting of one (1) group. The study will assess skin irritation as well as sensitization for d-ATS patch in healthy subjects. All three (3) articles (d-ATS patch, placebo patch, and saline patch) will be applied simultaneously on the back of each subject. Healthy subjects will be enrolled to participate in two (2) phases: A Screening Phase and a Treatment Phase. The total duration of the study for each subject will be about 10 - 16 weeks. The Re-challenge Test will only be performed for subjects who experience any type of sensitization during Challenge Period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject provides written informed consent prior to entering the study or undergoing any study procedures;
2. Healthy male and female (non-pregnant, non-lactating) 18 - 65 years of age inclusive;
3. Subject is considered by the Principal Investigator/Sponsor to be healthy on the basis of medical history, physical examination, vital signs, electrocardiogram (ECG) and clinical laboratory test results. Deviations or excursions considered to be non-clinically significant as per the Principal Investigator are acceptable;
4. Subject has a normal screening ECG; non-specific ST-T wave changes or other changes deemed by the Principal Investigator as not clinically significant are acceptable;
5. Female subject is (i) a woman physiologically incapable of becoming pregnant [confirmed to be post-menopausal (having amenorrhea for >12 months), has had a hysterectomy with or without bilateral oophorectomy at least 6 months prior to the Screening Visit] or (ii) a woman of childbearing potential (WOCBP) must have a negative pregnancy test at the Screening Visit and must agree to either abstain from sexual intercourse or use two forms of reliable barrier method of contraception (e.g., condom with spermicide, diaphragm, IUD, contraceptive sponge) for at least 14 days before and throughout the duration of study (from Screening Visit through the Follow-up Visit) or have used a hormonal method of contraception for at least 30 days before the study and will continue to use the same type of hormonal contraceptive during the study. Acceptable forms of birth control include (i) surgical sterilization (such as a tubal ligation), which occurred more than 3 months prior to the Screening Visit (ii) approved hormonal contraceptives (such as birth control pills, implants or injections), (iii) an intrauterine device, (iv) barrier method (condom or occlusive cap [diaphragm or cervical/vault caps] used with spermicidal foam/gel/film/cream/suppository), (v) Vasectomy in male partner, which occurred more than 3 months prior to the Screening Visit; bilateral oophorectomy may be enrolled. If the female subject agrees to use an occlusive cap/vault caps with spermicidal foam/gel/film/cream/suppository and her male partner agrees to use a condom with spermicidal foam/gel/film/cream/suppository, this would constitute as two methods of birth control;
6. Subject has a body mass index between 18 kg/m2 and 35 kg/m2, inclusive;
7. Subject has liver function tests such as alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase and bilirubin ≤1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%);
8. Subject is capable of understanding and complying with the protocol and has signed the Informed Consent Form.

Exclusion Criteria:

1. Subject is pregnant or lactating, or females planning a pregnancy during the course of the trial;
2. Subject with a history or presence of clinically significant disease (glaucoma, cardiovascular, hepatic, renal, gastrointestinal, neurologic, psychiatric, dermatologic, pulmonary, hematological, musculoskeletal, genitourinary, thromboembolic, advanced arteriosclerosis, hyperthyroidism, moderate to severe hypertension, asthma, urticaria, angioedema, edema, bronchospasm or immunologic disease or any other disorder). Conditions deemed not-clinically significant according to the Principal Investigator's discretion are acceptable;
3. Subject with a sitting blood pressure (BP) <90/50 or >139/89 mmHg and a sitting heart rate (HR) <45 or >90 beats/min;
4. Subject has a clinically significant ECG finding or QTcF interval >450 msec for males and >470 msec for females;
5. Subject has evidence of orthostatic hypotension (decrease of >20 mmHg systolic or >10 mmHg diastolic or both at supine for 5 minutes and again after assuming an upright position for 2 minutes) accompanied by symptoms (faintness, lightheadedness, dizziness, confusion);
6. Subject has a history of narcotic abuse, drug abuse, and alcoholism;
7. Subject has a clinically significant abnormal laboratory test result. Deviations considered to be non-clinically significant as per the Principal Investigator are acceptable;
8. Subject has a history of allergy or sensitivity to amphetamine or components in the patch;
9. Subject has a history or presence of significant skin disorder such as atopy, psoriasis, vitiligo, chronic cutaneous lupus erythematosus (CCLE), or conditions known to alter skin appearance (e.g., rash, infection, abnormally dry skin, abrasions), presence of tissue scar (e.g., tattoo) or excessive hair, body piercing, presence of open sores at the potential site of patch application or skin type that could, in any way, confound interpretation of the trial results (i.e., skin type VI on the Fitzpatrick scale);
10. Subject has a lifetime history of significant dermatologic cancers (e.g., melanoma, squamous cell carcinoma), except basal cell carcinomas that were superficial and did not involve the application sites;
11. Subject with any dermatologic diseases that might interfere with the evaluation of the test site reactions;
12. Subject has a history of any allergy to soaps, lotions, cosmetics, adhesives, or adhesive dressings;
13. Subject has a history of significant allergies (including food or drug allergies, minor seasonal allergies are allowed);
14. Subject with a history of a condition that would significantly influence the immune response (e.g., primary or acquired immunodeficiencies such as human immunodeficiency virus (HIV) positive or AIDS, allergic diseases such as anaphylaxis, asthma or generalized drug reaction, neoplasms such as lymphoma or leukemia, or rheumatoid arthritis);
15. Subject with a history of severe depression, psychoses, bipolar disorder, mania, aggression, marked anxiety, agitation, tension, seizures, Tourette's Syndrome, motor tics, glaucoma, migraines, or unexplained syncope;
16. Subject is on medications or treatments that would significantly influence or exaggerate responses to the test product or that would alter inflammatory or immune response to the product (e.g., cyclosporine, tacrolimus, systemic or topical corticosteroids, cytotoxic drugs, immune globulin, Bacillus Calmette-Guerin (BCG), monoclonal antibodies, radiation therapy) within 3 weeks prior to dosing;
17. Subject used any excluded over the counter medications (including herbal remedies) that would interfere with the objectives of the study or are contraindicated with the study drug for at least 7 days or 4-5 five half-lives, whichever is longer, prior to the first dose;
18. Subject used monoamine oxidase inhibitors within 14 days of dosing;
19. Subject used systemic or topical drugs and analgesics at the patch application site or antihistamines within 72 hours prior to dosing or systemic or topical corticosteroids within 3 weeks of study enrollment;
20. Subject with symptoms of significant acute illness at Screening or prior to dosing;
21. Subject with positive screen for hepatitis B and C;
22. Subject has been sunbathing, has used a tanning bed within 7 days of the Screening Visit or Admission, or has sunburn in the test area that could interfere with skin evaluation;
23. Subject who could foresee an intensive solar exposure during trial participation (UV radiation etc…) within 7 to 14 days of the Screening Visit;
24. Subject is a Study Investigator, Sub-Investigator, Study Coordinator or is employed by the site or the Sponsor, or is an immediate family member (e.g., spouse, parent, child or sibling, whether biological or legally adopted) of an employee of the site, participating Investigator, CRO or Sponsor;
25. Subject has received any investigational product or therapy within 30 days prior to study drug administration;
26. Any subject not able to meet study requirements in the opinion of the Principal Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-05-16 (Actual); Study Completion 2020-05-16 (Actual)

PRIMARY OUTCOMES:
Sensitization | 21 days
  Number of participants with sensitization potential after repeated exposure to d-ATS, placebo and saline patches in healthy adults
Irritation | 21 days
  Number of participants with skin irritation potential after repeated exposure to d-ATS, placebo and saline patches in healthy adults

CONTACTS AND LOCATIONS:
Overall Officials: George Harb, MD, Study Director — Noven Pharmaceuticals, Inc.
Locations (1):
- Noven Pharmaceuticals, Jersey City, New Jersey, United States